CLINICAL TRIAL: NCT02758522
Title: NPH and Regular Insulin in the Treatment of Inpatient Hyperglycemia: Comparison of 3 Basal-bolus Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. med. Hector Eloy Tamez Perez, Dr. med. Hector Eloy Tamez Perez, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MI13-005
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus; Hyperglycemia
Keywords: Diabetes Mellitus; Hospital Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Once-daily insulin (Active Comparator): 60% of total dose of insulin as NPH insulin in the once-daily regimen was administered subcutaneously before breakfast. Also, 40% in rapid insulin before meals (every 8 hours).
  Interventions: Drug: Once-daily Insulin
- Twice-daily insulin (Active Comparator): 60% of total dose of insulin as NPH insulin in the twice-daily regimen it was given before breakfast and before dinner. Also, 40% in rapid insulin before meals (every 8 hours).
  Interventions: Drug: Twice-daily Insulin
- Triple-daily insulin (Active Comparator): 60% of total dose of insulin as NPH insulin in the triple daily regimen it was administered before each meal. Also, 40% in rapid insulin before meals (every 8 hours).
  Interventions: Drug: Triple-daily Insulin

INTERVENTIONS:
Drug: Once-daily Insulin — Patients will receive NPH insulin in a once-daily regimen. The starting dose is calculate according to body mass index (BMI): 0.3 U/kg for BMI < 18 kg/m2, 0.4 U/kg for BMI 18-24.9 kg/m2, 0.5 U/kg for BMI 25-29.9 kg/m2 and 0.6 U/kg for BMI ≥ 30 kg/m2. The resulting dose will be fractioned to be given 60% as basal insulin (NPH) and 40% as prandial insulin (Regular). NPH insulin in the once-daily regimen will be administered subcutaneously before breakfast. Regular insulin subcutaneously wil be given in three equally divided doses before each meal.
  Arms: Once-daily insulin
Drug: Twice-daily Insulin — Patients receive NPH insulin in twice-daily regimen. The starting dose is calculated according to body mass index (BMI): 0.3 U/kg for BMI < 18 kg/m2, 0.4 U/kg for BMI 18-24.9 kg/m2, 0.5 U/kg for BMI 25-29.9 kg/m2 and 0.6 U/kg for BMI ≥ 30 kg/m2. The resulting dose will de fractioned to be given 60% as basal insulin (NPH) and 40% as prandial insulin (Regular). NPH insulin in the twice-daily regimen will be administered subcutaneously before breakfast and before dinner. Regular insulin will be given in three equally divided doses before each meal.
  Arms: Twice-daily insulin
Drug: Triple-daily Insulin — Patients receive NPH insulin in a triple-daily regimen. The starting dose was calculated according to body mass index (BMI): 0.3 U/kg for BMI < 18 kg/m2, 0.4 U/kg for BMI 18-24.9 kg/m2, 0.5 U/kg for BMI 25-29.9 kg/m2 and 0.6 U/kg for BMI ≥ 30 kg/m2. The resulting dose will be fractioned to be given 60% as basal insulin (NPH) and 40% as prandial insulin (Regular). NPH insulin in the triple daily regimen will be administered subcutaneously before each meal. Regular insulin will be given in three equally divided doses before each meal.
  Arms: Triple-daily insulin

SUMMARY:
The objective of this study is to compare the therapeutic efficacy of three regimens of insulin NPH/fast for optimal glycemic control in non-critical hospitalized patients.

DETAILED DESCRIPTION:
Patients will be randomly assigned to one of the three treatment regimens. Also, the use of oral antidiabetic drugs would be suspended during their stay at the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to medical services
* Persistent blood glucose level > 140 mg/dL
* With an expected stay ≥ 48 hours

Exclusion Criteria:

* Subjects with type 1 diabetes mellitus
* Parenteral nutrition
* Glucose levels ≥ 400 mg/dL at screening
* Diabetic ketoacidosis or non-ketosis hyperosmolar state
* Clinically relevant hepatic disease
* Glomerular filtration rate ≤ 30 ml/min
* Pregnancy
* Terminal disease
* Inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Glycemic control | Within the time the patient stays at hospital (2 to 14 days)
  The achievement of fasting glucose between 70-140 mg/dL and random glucose levels of <180 mg/dL

SECONDARY OUTCOMES:
Differences in the percentage of glucoses in the hypoglycemic range | Within the time the patient stays at hospital (2 to 14 days)
  Hypoglycemia was defined as glucose levels of < 70 mg/dL. Severe hypoglycemia was defined as glucose levels of < 40 mg/dL or the need of assistance.
Total insulin dose required during follow up and at discharge to achieve glycemic control | Within the time the patient stays at hospital (2 to 14 days)
Differences in hospital stay days | Within the time the patient stays at hospital (2 to 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Hector E Tamez-Perez, MD, PhD, Principal Investigator — Facultad de Medicina y Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Universidad Autonoma de Nuevo Leon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeSantis AJ, Schmeltz LR, Schmidt K, O'Shea-Mahler E, Rhee C, Wells A, Brandt S, Peterson S, Molitch ME. Inpatient management of hyperglycemia: the Northwestern experience. Endocr Pract. 2006 Sep-Oct;12(5):491-505. doi: 10.4158/EP.12.5.491. PMID 17002924
- [Background] Moghissi ES, Korytkowski MT, DiNardo M, Einhorn D, Hellman R, Hirsch IB, Inzucchi SE, Ismail-Beigi F, Kirkman MS, Umpierrez GE; American Association of Clinical Endocrinologists; American Diabetes Association. American Association of Clinical Endocrinologists and American Diabetes Association consensus statement on inpatient glycemic control. Diabetes Care. 2009 Jun;32(6):1119-31. doi: 10.2337/dc09-9029. Epub 2009 May 8. No abstract available. PMID 19429873
- [Background] Moghissi E. Hospital management of diabetes: beyond the sliding scale. Cleve Clin J Med. 2004 Oct;71(10):801-8. doi: 10.3949/ccjm.71.10.801. PMID 15529485
- [Background] Pichardo-Lowden AR, Fan CY, Gabbay RA. Management of hyperglycemia in the non-intensive care patient: featuring subcutaneous insulin protocols. Endocr Pract. 2011 Mar-Apr;17(2):249-60. doi: 10.4158/EP10220.RA. PMID 21041168
- [Background] Maynard G, Lee J, Phillips G, Fink E, Renvall M. Improved inpatient use of basal insulin, reduced hypoglycemia, and improved glycemic control: effect of structured subcutaneous insulin orders and an insulin management algorithm. J Hosp Med. 2009 Jan;4(1):3-15. doi: 10.1002/jhm.391. PMID 19140173
- [Background] Umpierrez GE, Smiley D, Zisman A, Prieto LM, Palacio A, Ceron M, Puig A, Mejia R. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes (RABBIT 2 trial). Diabetes Care. 2007 Sep;30(9):2181-6. doi: 10.2337/dc07-0295. Epub 2007 May 18. PMID 17513708
- [Background] ACE/ADA Task Force on Inpatient Diabetes. American College of Endocrinology and American Diabetes Association consensus statement on inpatient diabetes and glycemic control. Endocr Pract. 2006 Jul-Aug;12(4):458-68. doi: 10.4158/EP.12.4.458. No abstract available. PMID 16983798
- [Background] Mills RD, Schwartz F, Shubrook JH. Evaluation of diabetes management in a rural community hospital. Endocr Pract. 2008 Jan-Feb;14(1):50-5. doi: 10.4158/EP.14.1.50. PMID 18238741
- [Background] Schnipper JL, Ndumele CD, Liang CL, Pendergrass ML. Effects of a subcutaneous insulin protocol, clinical education, and computerized order set on the quality of inpatient management of hyperglycemia: results of a clinical trial. J Hosp Med. 2009 Jan;4(1):16-27. doi: 10.1002/jhm.385. PMID 19140191
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S64-71. doi: 10.2337/dc12-s064. No abstract available. PMID 22187472
- [Background] American Diabetes Association. Standards of medical care in diabetes--2012. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S11-63. doi: 10.2337/dc12-s011. No abstract available. PMID 22187469